CLINICAL TRIAL: NCT02957344
Title: Randomized Trial to Assess Parental Response to Different Presentations of Vaccination Data for Schools and Child Care Centers
Brief Title: Parental Views Related to Colorado State Legislation About Vaccinations, Schools, and Child Care Centers
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1149a
Record Dates: First submitted 2016-09-29; First posted 2016-11-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Children
Keywords: health communication; Zika virus; legislation; vaccination; Child Care
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Text without context
- Text with context
- Map without context
- Map with context

SUMMARY:
Through an online survey, participants will be shown different visual presentations of vaccination data related to schools and child care centers. Participants will rate how important this information is when thinking about their child's health and school choice. Participants will also be asked survey questions about their knowledge of Colorado state vaccination legislation, their opinions and practices related to childhood vaccinations, and their views of a Zika virus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* mother of a child 12 years of age or younger
* English literacy to complete the survey

Exclusion Criteria:

* respondent has a child of appropriate age but that child will not attend a school or child care center outside of the home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers of children 12 years of age or younger will be surveyed by email. They will be recruited from a group of women who have previously participated in a paper in-office survey at nine obstetrics/gynecology (OB/GYN) practices across the Front-Range region of Colorado. Women who completed the paper survey and provided contact information for future surveys may be contacted to participate in this survey.
Sampling Method: Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Survey/Questionnaire of parental knowledge and attitudes related to vaccines, schools, and child care centers. | On average within 2 months of survey invitation.
  Parental knowledge and attitudes will be evaluated related to legislation regarding schools and child care centers reporting vaccinations in Colorado. Survey is cross-sectional and will be administered to each participant once.

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No